CLINICAL TRIAL: NCT02858999
Title: Treatment of Primary Plasma Cell Leukaemia in Subjects Under the Age of 70: Phase II Multicentre Study
Brief Title: Treatment of Primary Plasma Cell Leukaemia in Subjects Under the Age of 70
Acronym: LPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOL09-DR-ROYER
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: primary plasma cell leukaemia; treatment
MeSH Terms: conditions — Multiple Myeloma

ARMS (1):
- treatment (Experimental): 12 weeks of induction chemotherapy by liposomal Bortezomib-Dexamethasone-Doxorubicin (PAD) alternating with Bortezomib-Dexamethasone-Cyclophosphamide (VCD) for a total of 4 cycles PAD-VCD
  Interventions: Drug: PAD-VCD

INTERVENTIONS:
Drug: PAD-VCD — 12 weeks of induction chemotherapy by liposomal Bortezomib-Dexamethasone-Doxorubicin (PAD) alternating with Bortezomib-Dexamethasone-Cyclophosphamide (VCD) for a total of 4 cycles

SUMMARY:
Plasma cell leukaemia is a rare variety of multiple myeloma with a poor prognosis. Plasma cell leukaemia is defined as: at least 2,000 circulating plasma cells per µL for a blood leukocyte count higher than 10,000/µL or 20% of plasma cells for a leukocyte count less than 10,000/µL. Plasma cell leukaemia can be either primary, when it constitutes the first manifestation of the disease, or secondary in the setting of relapsed/refractory multiple myeloma. Primary plasma cell leukaemia (PPL) is a rare disease, representing only 1 to 2% of all cases of multiple myelomas at diagnosis. As the annual incidence of multiple myeloma in France is about 4,000 new cases, an estimated 40 to 80 new cases of PPL would be observed each year.

Few data are currently available in the literature concerning the pathophysiology and therapeutic management of PPL, and are derived from retrospective series based small numbers of patients. The prognosis of PPL in response to conventional chemotherapy remains poor with a median survival of 7 to 14 months. However, longer survivals have been obtained with intensive therapy and haematopoietic stem cell transplantation (allogeneic or autologous HSCT).

The investigators propose to perform a prospective study of the management of patients with PPL under the age of 70 years, in combination with a laboratory study: 12 weeks of induction chemotherapy by liposomal Bortezomib-Dexamethasone-Doxorubicin (PAD) alternating with Bortezomib-Dexamethasone-Cyclophosphamide (VCD) for a total of 4 cycles. Peripheral blood stem cell collection after mobilization by G-CSF will be performed after high-dose Cyclophosphamide chemotherapy. Autologous HSCT conditioned by high-dose Melphalan will be performed during the following month for all responding patients. During the 3 months after this first autologous HSCT, allogeneic HSCT with attenuated conditioning will be proposed in patients under the age of 66 years in complete remission with a suitable donor, and another systematic autologous HSCT will be proposed in all other patients. For all patients not treated by allogeneic HSCT, consolidation/maintenance therapy will be performed 3 months after the second autologous HSCT: 4 quarterly consolidations with Bortezomib-Lenalidomide-Dexamethasone (VRD) with maintenance by 2 months of Lenalidomide between these cycles, for a total duration of one year.

The laboratory assessment will consist of blood and bone marrow samples systematically obtained at diagnosis for plasma cell phenotyping by cytometry, cytogenetics, FISH, study of the gene expression profile and SNParray. A DNA bank and plasma bank will be constituted. The investigators also propose to study residual disease by cytometry (after the first autologous HSCT, before and at the end of the consolidation/maintenance phase), as it increasingly appears to have a major impact on survival in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary plasma cell leukaemia corresponding to the International Myeloma Working Group definition.
* Patient not previously treated apart from a short course of corticosteroid therapy (dexamethasone 40 mg/day for 4 days).
* Age ≥ 18 years and < 70 years.
* Patient able to provide signed informed consent.
* Effective contraception when justified (oral contraception/protected intercourse).

Exclusion Criteria:

* Consent not obtained.
* Patient under judicial protection, or permanent or temporary guardianship.
* Previously treated multiple myeloma, secondary plasma cell leukaemia.
* ECOG performance status > 2.
* History of severe psychiatric illness, severe renal failure not attributable to PPL, heart failure (ejection fraction < 40%), bilirubin > 3N, transaminases or gamma GT > 4N.
* Peripheral neuropathy > NCI grade 2.
* Contraindication to high-dose corticosteroids, cyclophosphamide and anthracyclines.
* Hypersensitivity to bortezomib or lenalidomide.
* Pregnant woman or nursing mothers.
* Malignant disease except for basal cell carcinoma or cervical carcinoma in situ.
* Positive HIV serology; active hepatitis B or C.
* Participation in a clinical trial during the 60 days prior to inclusion.
* Patient not covered by French national health insurance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno ROYER, PhD, Principal Investigator — CHU Amiens
Locations (18):
- France (18):
  - CH Pays d'Aix, Aix-en-Provence
  - CHU Amiens, Amiens
  - CHU Besançon, Besançon
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CH Dunkerque, Dunkirk
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - AP-HP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Result] Royer B, Minvielle S, Diouf M, Roussel M, Karlin L, Hulin C, Arnulf B, Macro M, Cailleres S, Brion A, Brechignac S, Belhadj K, Chretien ML, Wetterwald M, Chaleteix C, Tiab M, Leleu X, Frenzel L, Garderet L, Choquet S, Fuzibet JG, Dauriac C, Forneker LM, Benboubker L, Facon T, Moreau P, Avet-Loiseau H, Marolleau JP. Bortezomib, Doxorubicin, Cyclophosphamide, Dexamethasone Induction Followed by Stem Cell Transplantation for Primary Plasma Cell Leukemia: A Prospective Phase II Study of the Intergroupe Francophone du Myelome. J Clin Oncol. 2016 Jun 20;34(18):2125-32. doi: 10.1200/JCO.2015.63.1929. Epub 2016 Apr 25. PMID 27114594